CLINICAL TRIAL: NCT02961764
Title: A Pragmatic Trial Designed to Evaluate a New Critical Pathway for Treatment of Patients With Acute Bacterial Skin and Skin Structure Infections
Brief Title: Evaluation of a New Critical Pathway for Treatment of Acute Bacterial Skin and Skin Structure Infections (ABSSSI)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMO-US-ID-0476
Record Dates: First submitted 2016-11-07; First posted 2016-11-11 (Estimated); Results first posted 2020-04-10 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-03

CONDITIONS: Acute Bacterial Skin and Skin Structure Infections
Keywords: Critical Pathways; Health Facilities; Clinical Protocols; Patient Satisfaction; Absenteeism; Anti-Bacterial Agents; Quality of Life; Economics, Medical; Health Resources; Health resource utilization; Acute bacterial skin and skin structure infection (ABSSSI)
MeSH Terms: conditions — Patient Satisfaction | interventions — dalbavancin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Usual Care (Active Comparator): Participants who receive Usual Care as prescribed by the physician as standard of care in clinical practice for the treatment of ABSSSI.
  Interventions: Drug: Usual Care
- New Critical Pathway (Active Comparator): The New Critical Pathway under study is defined as (1) use of guideline-based patient identification criteria, and, for those who meet these criteria, (2) use of dalbavancin, administered as a single intravenous (IV) dose of 1500 mg over 30 minutes for the treatment of ABSSSI.
  Interventions: Drug: Dalbavancin

INTERVENTIONS:
Drug: Usual Care — Usual care as prescribed by the physician as standard of care in clinical practice for the treatment of ABSSSI.
  Arms: Usual Care
Drug: Dalbavancin — Dalbavancin administered as a single IV dose of 1500 mg over 30 minutes.
  Other Names: Dalvance®
  Arms: New Critical Pathway

SUMMARY:
This study will evaluate a new critical pathway (use of guideline-based patient identification criteria and for those who meet these criteria, use of dalbavancin) for the treatment of ABSSSI compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

* Presents to the Emergency Department (ED) and meets the clinical definition for Acute Bacterial Skin and Skin Structure Infections (ABSSSI)
* Known or suspected gram-positive infection.

Exclusion Criteria:

* Known or suspected gram-negative infections, anaerobic infections, or fungemia
* Known or suspected infections that are severe, life threatening or are not included in the ABSSSI Food and Drug Administration (FDA) guidance
* Injection drug users with a fever
* Severe neurological disorder leading to immobility or confined to a wheelchair
* Bilateral Lower extremity involvement of the suspected infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2016-11-29 (Actual); Primary Completion 2019-03-29 (Actual); Study Completion 2019-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Gillard, Study Director — Allergan
Locations (11):
- United States (11):
  - Maricopa Medical Center, Phoenix, Arizona
  - Olive View-UCLA Medical Center, Sylmar, California
  - Hartford Hospital, Hartford, Connecticut
  - Tampa General Hospital, Tampa, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Johns Hopkins Hospital, Baltimore, Maryland
  - University of Massachusetts, Worcester, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Wayne State University, Detroit, Michigan
  - ProMedica Monroe Regional Hospital, Monroe, Michigan
  - Truman Medical Centers, Kansas City, Missouri

REFERENCES:
- [Derived] Talan DA, Mower WR, Lovecchio FA, Rothman RE, Steele MT, Keyloun K, Gillard P, Copp R, Moran GJ. Pathway with single-dose long-acting intravenous antibiotic reduces emergency department hospitalizations of patients with skin infections. Acad Emerg Med. 2021 Oct;28(10):1108-1117. doi: 10.1111/acem.14258. Epub 2021 May 5. PMID 33780567
- See also: More Information — http://allerganclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Care | New Critical Pathway
Started | 160 | 153
Completed | 121 | 128
Not Completed | 39 | 25
Not completed — Protocol Violation | 0 | 1
Not completed — Death | 2 | 0
Not completed — Lost to Follow-up | 35 | 24
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) population consists of all enrolled patients that has received at least one dose of antibiotics or one dose of dalbavancin for inclusion.
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | New Critical Pathway | Total
Number analyzed (Participants) | 156 | 153 | 309
Age, Customized [Count of Participants; unit: Participants]
  <20 years | 1 | 2 | 3
  20-29 years | 28 | 14 | 42
  30-39 years | 31 | 40 | 71
  40-49 years | 25 | 29 | 54
  50-59 years | 37 | 31 | 68
  60-69 years | 22 | 24 | 46
  70-79 years | 8 | 9 | 17
  80-89 years | 3 | 3 | 6
  90-98 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 54 | 110
  Male | 100 | 99 | 199
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 39 | 43 | 82
  Not Hispanic or Latino | 116 | 107 | 223
  Unknown or Not Reported | 1 | 3 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White or Caucasian | 89 | 91 | 180
  Black or African American | 30 | 39 | 69
  American Indian or Alaska Native | 6 | 2 | 8
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Other | 17 | 16 | 33
  Patient chose not to answer | 13 | 3 | 16

OUTCOME MEASURES:

1. Primary Outcome: Hospital Admission Rate at Initial Episode of Care
Time Frame: 44 Days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 156 | 153
Participants
  Yes | 60 | 27
  No | 96 | 126
Statistical Analysis 1: Comparison: Usual Care vs New Critical Pathway; Test type: Superiority; p < 0.001, Fisher Exact; Odds Ratio (OR) = 0.289, 95% CI 2-sided [0.156 to 0.532]

2. Secondary Outcome: Number of Total Admitted Hospital Days
Description: Number of days during the initial hospitalization (for those initially hospitalized) and all other hospitalizations
Time Frame: 44 Days
Population: FAS population consists of all enrolled patients that has received at least one dose of antibiotics or one dose of dalbavancin for inclusion. Patients who discontinued prior to day 14 of the study were excluded from the Follow-up and Entire Study Duration analyses due to missing data for 15-44 day period.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 145 | 141
Days | 2.3 (3.74) | 1.2 (2.58)
Statistical Analysis 1: Comparison: Usual Care vs New Critical Pathway; Test type: Superiority; p = 0.005, t-test, 1 sided

3. Secondary Outcome: Total Length of Stay in Emergency Department (ED) During the Initial Episode of Care
Description: Time spent in ED in hours from triage to release (either admitted to the hospital, admitted to observation, or released to home)
Time Frame: Initial Care: 14 Days
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 156 | 153
Hours | 7.7 (9.09) | 6.1 (3.94)
Statistical Analysis 1: Comparison: Usual Care vs New Critical Pathway; Test type: Superiority; p = 0.050, t-test, 1 sided

4. Secondary Outcome: Number of Participants With Infection-related Major Surgical Interventions That Required Operating Room Time
Description: Number of all major surgical interventions unexpected or expected that required operating room time
Time Frame: 44 Days
Population: Full analysis set (FAS) population consists of all enrolled patients that has received at least one dose of antibiotics or one dose of dalbavancin for inclusion. Patients who discontinued prior to day 14 of the study were excluded from the Follow-up and Entire Study Duration analyses due to missing data for 15-44 day period.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 145 | 141
Participants
  No Surgeries | 107 | 106
  Any Surgeries | 38 | 35

5. Secondary Outcome: Number of Infection-related Total Admitted Hospital Days
Time Frame: 44 Days
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 145 | 141
Days | 2.0 (3.06) | 1.0 (2.36)
Statistical Analysis 1: Comparison: Usual Care vs New Critical Pathway; Test type: Superiority; p = 0.002, t-test, 1 sided

6. Secondary Outcome: Number of Participants With Infection-related Hospitalizations
Description: Number of days of hospitalization during the initial hospitalization (for those initially hospitalized) and all other infection-related hospitalizations
Time Frame: 44 Days
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 145 | 141
Participants
  None | 85 | 110
  Any | 60 | 31

7. Secondary Outcome: Number of Participants With Infection-related Hospitalizations During Initial Care and Follow-up That Resulted in Admission to Intensive Care Unit
Time Frame: 44 Days
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 145 | 141
Participants
  Admission to ICU | 3 | 0

8. Secondary Outcome: Number of Participants With All Cause Hospitalizations in the 30 Days Post Discharge From the Hospital or Release From the ED
Time Frame: Follow-up: 30 Days
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 145 | 141
Participants | 7 | 12

9. Secondary Outcome: Number of Participants With Infection-related Emergency Department (ED) Visits
Time Frame: 44 Days
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 145 | 141
Participants | 22 | 19

10. Secondary Outcome: Number of Participants With Infection-related Outpatient Healthcare Visits
Time Frame: 44 Days
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 145 | 141
Participants | 57 | 39

11. Secondary Outcome: Use of a Peripherally-Inserted Central Catheter (PICC) Line or Central Line to Administer Antibiotic Therapy
Time Frame: 44 Days
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 145 | 141
Participants
  Peripheral IV | 93 | 141
  Central line | 0 | 0
  PICC line | 1 | 1
  No Line | 143 | 136

12. Secondary Outcome: Number of Participants With Infection-related Healthcare Visits Due to PICC Line or Central Line Used to Administer Antibiotic Therapy
Time Frame: 44 Days
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 145 | 141
Participants
  1 occurence | 2 | 1

13. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Time Frame: 44 Days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 156 | 153
Participants | 11 | 16

14. Secondary Outcome: Patient Satisfaction With Care: Overall Health
Description: Patient satisfaction with care as assessed through the ABSSSI Patient Satisfaction Survey (patient reported).
Time Frame: Day 14
Population: FAS population. 119 and 124 patients provided any survey data in the usual care group and the new critical pathway group, respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 119 | 124
Participants
  Excellent | 12 | 22
  Very good | 38 | 31
  Good | 35 | 40
  Fair | 30 | 23
  Poor | 4 | 8

15. Secondary Outcome: Patient Satisfaction With Care: Wait in Emergency Room
Description: Patients rated their satisfaction on a 10-point scale, where 0 was the worst experience possible and 10 the best experience possible.
Time Frame: Day 14
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 119 | 124
scores on a scale | 7.8 (2.63) | 8.3 (2.25)

16. Secondary Outcome: Patient Satisfaction With Care: Hospitalization
Description: Patient satisfaction with care as assessed through the ABSSSI Patient Satisfaction Survey (patient reported).
Time Frame: Day 14
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 119 | 124
Participants
  Yes | 63 | 27
  No | 56 | 97

17. Secondary Outcome: Patient Satisfaction With Care: Satisfaction With Hospital Stay
Description: as for outcome 15
Time Frame: Day 14
Population: FAS population. 119 and 124 patients provided any survey data in the usual care group and the new critical pathway group, respectively. 63 and 27 patients had a hospital stay in the usual care group and new critical pathway group, respectively.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 63 | 27
Scores on a Scale | 8.2 (2.19) | 8.0 (1.85)

18. Secondary Outcome: Patient Satisfaction With Care: Factors for Dissatisfaction With Your Hospital Stay
Description: Patient satisfaction with care as assessed through the ABSSSI Patient Satisfaction Survey (patient reported).
Time Frame: Day 14
Population: FAS population. 119 and 124 patients provided any survey data in the usual care group and the new critical pathway group, respectively. Patients may have checked multiple responses.
Measure: Number; unit: Participant
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 119 | 124
Participant
  Hospital stay interfered with work/school | 11 | 8
  Stay got in way of daily normal activities | 11 | 10
  Stay got in the way of providing care to others | 8 | 8
  Hospital stay was expensive | 2 | 6
  Did not provide adequate monitoring by providers | 3 | 1
  Did not provide well trained healthcare providers | 3 | 0
  Hospital stay made me feel worse | 3 | 0
  Hospital stay made me feel concerned | 14 | 7
  Hospital stay was uncomfortable | 11 | 5
  Hospital stay disrupted my sleep | 12 | 6
  Other | 7 | 2
  I was not dissatisfied with my hospital stay | 33 | 12

19. Secondary Outcome: Patient Satisfaction With Care: Received IV Antibiotic Therapy for Skin Infections
Description: Patient satisfaction with care as assessed through the ABSSSI Patient Satisfaction Survey (patient reported).
Time Frame: Day 14
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 119 | 124
Participants
  Yes | 87 | 119
  No | 32 | 5

20. Secondary Outcome: Patient Satisfaction With Care: Satisfaction With Receiving IV Antibiotic Therapy
Description: as for outcome 15
Time Frame: Day 14
Population: 119 & 124 patients provided any survey data in the usual care group & new critical pathway group; 87 & 119 patients received IV antibiotic therapy in the usual care group & new critical pathway group; 86 and 119 patients answered this question in the usual care group & new critical pathway group, respectively.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 86 | 119
Scores on a Scale | 8.7 (2.16) | 9.0 (1.63)

21. Secondary Outcome: Patient Satisfaction With Care: Factors Contributing to Satisfaction With Receiving IV
Description: Patient satisfaction with care as assessed through the ABSSSI Patient Satisfaction Survey (patient reported).
Time Frame: Day 14
Population: as for outcome 18
Measure: Number; unit: Participants
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 119 | 124
Participants
  Allowed me to return to work/school | 37 | 50
  Allowed me to return to daily normal activities | 48 | 81
  Allowed me to return to providing care to others | 38 | 52
  IV antibiotic therapy was affordable | 29 | 45
  Administered at appointments that I could schedule | 4 | 11
  Administered quickly once arrived at appt | 4 | 17
  Administered at setting that had convenient hours | 3 | 16
  Ensured regular monitoring by healthcare providers | 26 | 29
  Administered by skilled healthcare providers | 51 | 58
  IV antibiotic therapy made me feel better | 55 | 80
  Allowed to receive care for skin infection at home | 4 | 10
  Convenient to administer by self/caregiver at home | 2 | 4
  Other | 4 | 8
  Not satisfied with receiving IV antibiotic therapy | 9 | 3

22. Secondary Outcome: Patient Satisfaction With Care: Factors Contributing to Dissatisfaction With Receiving IV
Description: Patient satisfaction with care as assessed through the ABSSSI Patient Satisfaction Survey (patient reported).
Time Frame: 14 Days
Population: as for outcome 18
Measure: Number; unit: Participants
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 119 | 124
Participants
  Got in the way of work/school | 2 | 1
  Got in way of performing daily normal activities | 3 | 4
  Got in the way of providing care to others | 1 | 1
  IV antibiotic therapy was expensive | 0 | 0
  Required me to make appointments | 1 | 0
  Administered at healthcare setting w/limited hours | 1 | 0
  Required traveling to and from appointments | 0 | 0
  Required to wait to be seen by provider | 1 | 2
  IV antibiotic therapy took too long to administer | 1 | 3
  Required having a PICC or central line inserted | 2 | 2
  Caused an IV site infection | 0 | 0
  IV antibiotic therapy made me feel worse | 2 | 2
  Not adequately monitored by healthcare providers | 1 | 0
  Not administered by skilled healthcare providers | 1 | 0
  IV antibiotic therapy made me feel concerned | 2 | 2
  Required a nurse/healthcare worker coming to home | 0 | 0
  Required administration to self/caregiver at home | 0 | 0
  Other | 4 | 1
  Not dissatisfied w/receiving IV antibiotic therapy | 72 | 105

23. Secondary Outcome: Patient Satisfaction With Care: IV Therapy Hindering Normal Activities of Daily Living
Description: Patient satisfaction with care as assessed through the ABSSSI Patient Satisfaction Survey (patient reported).
Time Frame: Day 14
Population: 119 & 124 patients provided any survey data in the usual care group & new critical pathway group; 87 & 119 patients received IV antibiotic therapy in the usual care group & new critical pathway group; 87 and 118 patients answered this question in the usual care group & new critical pathway group, respectively
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 87 | 118
Participants
  None of the time | 66 | 94
  A little of the time | 6 | 10
  Some of the time | 6 | 11
  Most of the time | 5 | 1
  All of the time | 4 | 2

24. Secondary Outcome: Patient Satisfaction With Care: Concerned About Receiving Your IV Therapy
Description: Patient satisfaction with care as assessed through the ABSSSI Patient Satisfaction Survey (patient reported).
Time Frame: Day 14
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 87 | 118
Participants
  None of the time | 62 | 80
  A little of the time | 8 | 19
  Some of the time | 8 | 12
  Most of the time | 5 | 3
  All of the time | 4 | 4

25. Secondary Outcome: Patient Satisfaction With Care: Satisfied With the Number of IV Infusions Received Per Day
Description: as for outcome 15
Time Frame: Day 14
Population: 119 & 124 patients provided any survey data in the usual care group & new critical pathway group; 87 & 119 patients received IV antibiotic therapy in the usual care group & new critical pathway group; 85 and 118 patients answered this question in the usual care group & new critical pathway group, respectively
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 85 | 118
Scores on a scale | 8.4 (2.36) | 9.0 (1.70)

26. Secondary Outcome: Patient Satisfaction With Care: Satisfaction With the Average Time to Administer Each IV
Description: as for outcome 15
Time Frame: Day 14
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 85 | 118
Scores on a Scale | 8.6 (1.87) | 8.8 (1.88)

27. Secondary Outcome: Patient Satisfaction With Care: Time to Travel to Appointments to Receive IV
Description: Patient satisfaction with care as assessed through the ABSSSI Patient Satisfaction Survey (patient reported).
Time Frame: 14 days
Population: 119 & 124 patients provided any survey data in the usual care group & new critical pathway group; 87 & 119 patients received IV antibiotic therapy in the usual care group & new critical pathway group; 86 and 118 patients answered this question in the usual care group & new critical pathway group, respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 86 | 118
Participants
  Less than 15 minutes | 7 | 19
  16 - 30 minutes | 5 | 17
  31 - 60 minutes | 2 | 4
  61 - 90 minutes | 1 | 1
  More than 90 minutes | 2 | 0
  I did not need to travel to my appointments | 68 | 77
  I don't remember | 1 | 0

28. Secondary Outcome: Patient Satisfaction With Care: Average Time to be Seen by a Healthcare Provider
Description: Patient satisfaction with care as assessed through the ABSSSI Patient Satisfaction Survey (patient reported).
Time Frame: 14 days
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 86 | 118
Participants
  Less than 15 minutes | 4 | 17
  16 - 30 minutes | 7 | 10
  31 - 60 minutes | 3 | 4
  61 - 90 minutes | 3 | 2
  More than 90 minutes | 2 | 8
  I did not need to wait for my appointments | 67 | 75
  I don't remember | 0 | 2

29. Secondary Outcome: Patient Satisfaction With Care: Healthcare Setting Preferred if Treated Again for a Skin Infection With IV
Description: Patient satisfaction with care as assessed through the ABSSSI Patient Satisfaction Survey (patient reported).
Time Frame: 14 Days
Population: FAS population. 119 and 124 patients provided any survey data in the usual care group and the new critical pathway group; 116 and 123 patients answered this question in the usual care group & new critical pathway group, respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 116 | 123
Participants
  Overnight hospital stay for one or more nights | 42 | 17
  Outpatient care: Brief hospital visit w/no stay | 74 | 106

30. Secondary Outcome: Patient Satisfaction With Care: Factors Contributing to Preference for Outpatient Care
Description: Patient satisfaction with care as assessed through the ABSSSI Patient Satisfaction Survey (patient reported).
Time Frame: 14 Days
Population: as for outcome 18
Measure: Number; unit: Participants
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 119 | 124
Participants
  To avoid hospital stay for 1 or more nights | 52 | 91
  To allow me to return to work/school | 37 | 44
  To return to performing daily normal living | 48 | 65
  To allow me to return to providing care to others | 27 | 36
  Outpatient care would be more affordable | 21 | 38
  Outpatient care would be more convenient | 43 | 64
  To ensure monitoring by healthcare providers | 10 | 22
  Administered by skilled healthcare providers | 17 | 27
  Other | 3 | 1
  I would not prefer outpatient care | 38 | 14

31. Secondary Outcome: Patient Satisfaction With Care: Regimen Preferred if Treated Again for a Similar Skin Infection With IV
Description: Patient satisfaction with care as assessed through the ABSSSI Patient Satisfaction Survey (patient reported).
Time Frame: Day 14
Population: FAS population. 119 and 124 patients provided any survey data in the usual care group and the new critical pathway group; 117 and 121 patients answered this survey question in the usual care group & new critical pathway group, respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 117 | 121
Participants
  Regimen 1 | 65 | 107
  Regimen 2 | 14 | 6
  Regimen 3 | 38 | 8

32. Secondary Outcome: Patient Satisfaction With Care: Time Willing to Spend Receiving Each IV
Description: Patient satisfaction with care as assessed through the ABSSSI Patient Satisfaction Survey (patient reported).
Time Frame: Day 14
Population: FAS population. 119 and 124 patients provided any survey data in the usual care group and the new critical pathway group; 117 and 123 patients answered this survey question in the usual care group & new critical pathway group, respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 117 | 123
Participants
  About 30 minutes or less | 73 | 87
  About 1 hour | 28 | 32
  About 1.5 to 2 hours | 13 | 3
  About 3 hours or longer | 3 | 1

33. Secondary Outcome: Patient Satisfaction With Care: Find Value in a Physician
Description: Patient satisfaction with care as assessed through the ABSSSI Patient Satisfaction Survey (patient reported).
Time Frame: Day 14
Population: FAS population. 119 and 124 patients provided any survey data in the usual care group and the new critical pathway group; 115 and 123 patients answered this survey question in the usual care group & new critical pathway group, respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 115 | 123
Participants
  Definitely not | 13 | 5
  Probably not | 13 | 8
  Probably so | 38 | 37
  Definitely so | 51 | 73

34. Secondary Outcome: Patient Work and Productivity Loss as Assessed Through the Work Productivity and Activity Impairment Questionnaire
Description: Number of days with lost/reduced productivity during follow-up, as measured with Work Productivity and Activity Impairment (WPAI) Questionnaire
Time Frame: Day 14
Population: FAS population. 119 and 123 patients provided any survey data in the usual care group and the new critical pathway group; 53 and 48 patients completed all survey questions in the usual care group and new critical pathway group, respectively. 61 and 56 were employed.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 119 | 123
Percentage
  Absenteeism: number analyzed (Participants) | 58 | 54
  Absenteeism | 17.4 (31.96) | 18.9 (33.49)
  Impairment while working: number analyzed (Participants) | 53 | 48
  Impairment while working | 14.5 (24.14) | 10.8 (22.30)
  Overall work impairment: number analyzed (Participants) | 53 | 48
  Overall work impairment | 21.3 (29.04) | 16.4 (26.82)
  Activity impairment | 24.2 (34.06) | 15.9 (28.88)

35. Secondary Outcome: Patient Health-related Quality of Life (HRQoL) Assessed by the Short Form 12 (SF-12) 12-Item Patient Questionnaire
Description: The SF-12 yields a physical and a mental health component summary score (referred to as physical component summary score [PCS] and mental component summary score [MCS]). The PCS and MCS follow a t-score distribution, i.e. mean of 50 and standard deviation of 10 in the general US population, meaning all scores above or below 50 are above and below the average, respectively, in the US general population.
Time Frame: Day 14
Population: FAS population. 119 and 122 patients provided any and all survey data in the usual care group and the new critical pathway group, respectively.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 119 | 122
Score on a Scale
  Mental Health Component Score | 51.2 (10.36) | 52.6 (9.63)
  Physical Health Component Score | 46.4 (10.36) | 47.8 (9.39)

ADVERSE EVENTS:
Time Frame: Adverse events were collected up to 44 days. Initial care is the date of enrollment to 10-14 days and follow-up is 30 days after initial care.
Arm/Group | Usual Care | New Critical Pathway
All-Cause Mortality (participants affected / at risk) | 2/156 | 2/153
Serious Adverse Events (participants affected / at risk) | 11/156 | 16/153
Other Adverse Events (participants affected / at risk) | 4/156 | 16/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Usual Care (N=156) | New Critical Pathway (N=153)
CELLULITIS (Infections and infestations) | 2 | 8
SKIN INFECTION (Infections and infestations) | 2 | 0
BRONCHITIS (Infections and infestations) | 1 | 0
ABSCESS (Infections and infestations) | 0 | 1
BACTERAEMIA (Infections and infestations) | 0 | 1
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 0 | 1
LYMPHANGITIS (Infections and infestations) | 0 | 1
SKIN BACTERIAL INFECTION (Infections and infestations) | 0 | 1
SUBCUTANEOUS ABSCESS (Infections and infestations) | 0 | 1
TREATMENT FAILURE (General disorders) | 2 | 0
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 | 0
ANAPHYLACTIC REACTION (Immune system disorders) | 1 | 0
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 | 0
SOFT TISSUE INJURY (Injury, poisoning and procedural complications) | 0 | 1
BLOOD CULTURE POSITIVE (Investigations) | 1 | 0
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 | 0
ECTOPIC PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 1 | 0
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 0 | 1
HIDRADENITIS (Skin and subcutaneous tissue disorders) | 0 | 1
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 0 | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Usual Care (N=156) | New Critical Pathway (N=153)
Diarrhoea (Gastrointestinal disorders) | 2 | 8
Cellulitis (Infections and infestations) | 2 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2018-01-11): https://cdn.clinicaltrials.gov/large-docs/64/NCT02961764/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-05): https://cdn.clinicaltrials.gov/large-docs/64/NCT02961764/SAP_001.pdf